CLINICAL TRIAL: NCT01594008
Title: Does Blueberry Intake Alleviate Postprandial Lipemia-induced Inflammation?
Brief Title: The Effects of Antioxidants in Blueberry Powder on Inflammation Induced by a Single High Fat Meal.
Acronym: FL89
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: U.S. Highbush Blueberry Council (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 250305-3
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2013-05

CONDITIONS: Inflammation
Keywords: Toll like receptors; Inflammation; Anthocyanins; Blueberries
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Breakfast meal with placebo powder — Zero serving equivalents (1 serving equivalent = ½ cup fresh raw blueberries) of blueberries in the form of a mixed side dish comprising frozen yogurt, sugar, and placebo powder.
Other: Breakfast meal with 2 serving equivalents of blueberries — Two serving equivalents (1 serving equivalent = ½ cup fresh raw blueberries) of blueberries in the form of a mixed side dish comprising frozen yogurt, sugar, and freeze-dried blueberry powder.
Other: Breakfast meal with 4 serving equivalents of blueberries — Four serving equivalents (1 serving equivalent = ½ cup fresh raw blueberries) of blueberries in the form of a mixed side dish comprising frozen yogurt, sugar, and freeze-dried blueberry powder.

SUMMARY:
The goal of the study is to find out whether a high fat meal increases blood lipids and causes monocyte (white blood cell) activation, and whether blueberry intake at the same meal lessens monocyte activation in healthy people.

DETAILED DESCRIPTION:
This study was designed as a single blind, placebo-controlled crossover study. Subjects were never told what dose of blueberry powder was given. Researchers handling samples and data did not know what dose of blueberry powder subjects received on test day 2 or 3. The frozen blueberry yogurt supplemented with either control or blueberry powder was coded by letter, and samples were coded by test day: since the control powder was given on the first day to all subjects, the laboratory staff analyzing the samples would have known that the first day samples were from the subjects receiving the control powder.The provision of the control powder on the first day to all subjects was done to mitigate potential carry over effects of the blueberry powder.The randomization plan for the two doses (two vs four servings) of blueberry powder was uploaded into a spreadsheet of which only the registered dietitian, the Human Studies Manager, and the Metabolic Kitchen and Human Feeding Laboratory staff had access. Subjects were instructed by a registered dietitian to follow a low polyphenol and omega-3 diet and limit consumption of fruits, vegetables, soy, fatty fish (e.g. salmon), whole grains, nuts, coffee, tea, and chocolate starting 3 days prior to each test day. The night before each test day, subjects were required to eat a standardized dinner provided by the WHNRC. Since a previous meal may impact the postprandial response of the next, subjects were fed a dinner that consisted of a burrito with tortilla, chicken, cheese, oil, and pinto beans as well as yogurt and lemonade. On each test day, subjects arrived at the WHNRC after a 12-hour overnight fast. Subjects had their body temperature, blood pressure, and weight measured, and then had blood withdrawn. Subjects were fed the MHF breakfast supplemented with a frozen yogurt containing either control or blueberry powder. Subjects were given 20 minutes to consume the entire breakfast. Subjects were instructed not to eat or drink anything other than plain water. Three and one-half hours following consumption of the test meal each subject returned to the WHNRC for a postprandial blood draw. Postprandial hypertriglyceridemia peaks on average 3.5 hours after the consumption of a high fat breakfast, thus the 3.5 hour blood draw provides the highest concentration of TGRL. Subjects were allowed to return to their normal activities after the morning meal before the postprandial blood draw. Following the postprandial blood draw, subjects were allowed to return to their normal dietary habits until three days prior to their next test day. Subjects were fed the control powder on their first test day. On the second and third test days subjects were fed varying amounts of the blueberry powder that were equivalent to two or four servings of fresh blueberries (24.1 g and 48.2 g of blueberry powder, respectively) in a random order.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Able to complete study procedures
* Body Mass Index 18 - 24.9 kg/m2

Exclusion Criteria:

* Diabetes mellitus
* Kidney disease
* Liver disease
* Thyroid disease
* Bleeding disorders
* Autoimmune diseases and other inflammatory disease
* Cancer, unless in remission for > 5 years
* Blood cell counts outside the normal range for age and gender
* Blood chemistry panels outside the normal range for age and gender
* Blood cholesterol greater than 240 mg/dL
* Blood triacylglycerol greater than 300 mg/dL
* Hemoglobin less than 11.5 g/dL
* Hypertension, blood pressure greater than 140/90 mmHg
* Follow a vegetarian diet
* Smoke or use tobacco products
* Drink more than one alcoholic beverage per day
* Taking cholesterol-lowering or blood pressure medication
* Daily or regular use of antihistamines
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs)
* Use of steroids for asthma or other inflammatory diseases
* Use of thyroid-regulating drugs
* Use of over the counter weight loss products
* Known allergies or sensitivities to food ingredients in the test meals
* Taking fish or algal oil supplements and unwilling to stop
* Pregnant and lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Monocyte activation in whole blood | Change in activation from 0 to 3.5 hours
  Monocyte activation assay in whole blood will be measured by IL-1Beta secretion and other cytokines (TNF-alpha, INFγ).

SECONDARY OUTCOMES:
Peripheral blood mononuclear (PBMC) activation | Change from 0 to 3.5 hours
  Peripheral blood mononuclear (PBMC) activation in response to autologous fasting and postprandial serum will be analyzed for IL-1beta secretion and other cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hwang, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center; John Rutledge, MD, Principal Investigator — University of California, Davis
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Derived] Ono-Moore KD, Snodgrass RG, Huang S, Singh S, Freytag TL, Burnett DJ, Bonnel EL, Woodhouse LR, Zunino SJ, Peerson JM, Lee JY, Rutledge JC, Hwang DH. Postprandial Inflammatory Responses and Free Fatty Acids in Plasma of Adults Who Consumed a Moderately High-Fat Breakfast with and without Blueberry Powder in a Randomized Placebo-Controlled Trial. J Nutr. 2016 Jul;146(7):1411-9. doi: 10.3945/jn.115.223909. Epub 2016 Jun 15. PMID 27306892
- See also: USDA Western Human Nutrition Research Center — http://www.ars.usda.gov/Main/docs.htm?docid=11240